CLINICAL TRIAL: NCT02160132
Title: Effect and Security of Steroids Therapy for Patients of IgA Nephropathy With Active Pathological Changes : A Prospective, Randomized, Controlled, Multi-Center Clinical Trial.
Brief Title: A Controlled Study of Steroids Therapy for Patients of IgA Nephropathy With Active Pathological Changes.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, The Sixth Affiliated Hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usix-IgAN-001
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Glomerulonephritis, IGA; Peripapillary Crescent; Necrosis; Steroid Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1-2-3Group (Experimental): Methylprednisolone 0.5g/d intravenously for 3 consecutive days in the 1st-2nd-3rd month ,and oral methylprednisolone 0.4mg/kg/d on consecutive days for 6 months.
  Interventions: Drug: Methylprednisolone(intravenously in the 1st-2nd-3rd month )
- B 1-3-5Group (Active Comparator): Methylprednisolone 0.5g/d intravenously for 3 consecutive days in the 1st-3rd-5th month ,and oral methylprednisolone 0.4mg/kg/d on consecutive days for 6 months.
  Interventions: Drug: Methylprednisolone(intravenously in the 1st-3rd-5th month)

INTERVENTIONS:
Drug: Methylprednisolone(intravenously in the 1st-2nd-3rd month ) — Methylprednisolone 0.5g/d intravenously for 3 consecutive days in the 1st-2nd-3rd month ,and oral methylprednisolone 0.4mg/kg/d on consecutive days for 6 months.
  Arms: A 1-2-3Group
Drug: Methylprednisolone(intravenously in the 1st-3rd-5th month) — Methylprednisolone 0.5g/d intravenously for 3 consecutive days in the 1st-3rd-5th month ,and oral methylprednisolone 0.4mg/kg/d on consecutive days for 6 months.
  Arms: B 1-3-5Group

SUMMARY:
This prospective, randomized, controlled, multi-center clinical trial will evaluate the effect and security of steroids therapy for patients of IgA nephropathy with active pathological changes,including crescents,necrosis and microthrombus.

DETAILED DESCRIPTION:
It has been reported that for urinary protein excretion that is persistently more than 1g/24h and eGFR>50ml/min/1.73m2 in IgA nephropathy(IgAN), the KDIGO guidelines suggest a 6-month course of glucocorticoids. The famous study by Pozzi C has proved that for patients of IgAN with proteinuria of 1.0-3.5g/24h and serum creatinine concentrations of 133 umol/L or less, a 6-month course of steroid treatment(1g/d methylprednisolone intravenously for 3 consecutive days,with the course repeated 2 months and 4 months later,then oral prednisone 0.5mg/kg/d on alternate days for 6 months) could significantly reduce proteinuria and protect against renal function deterioration in IgAN. Furthermore, as we know, active pathological changes in IgAN,including crescents,necrosis and microthrombus,which may turn fibrosis after three months would effect the prognosis.This will be a prospective, randomized, controlled, multi-center study. Patients in treatment group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-2nd-3rd month ,then oral methylprednisolone 0.4mg/kg/d on consecutive days Patients in control group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-3rd-5th month ,then oral methylprednisolone 0.4mg/kg/d on consecutive days. After followed-up for 6 months, the curative effect of steroid therapy on proteinuria and the progression of IgAN will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 14~65 years, regardless of gender
* Clinical evaluation and renal biopsy diagnostic for IgA nephropathy, presenting with active pathological changes,including cellular crescents,necrosis and microthrombus.
* Average urinary protein excretion of 0.5~3.5g/24h on two successive examinations.
* eGFR ≥ 50 ml/min/1.73 m2
* Willingness to sign an informed consent.

Exclusion Criteria:

* Secondary IgAN such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B -associated nephritis.
* Rapidly progressive nephritic syndrome (crescent formation≥50%).
* Acute renal failure, including rapidly progressive IgAN.
* Current or recent (within 30 days) exposure to high-dose of steroids or immunosuppressive therapy (CTX、MMF、CsA、FK506).
* Date of renal biopsy exceeds more than 30 days.
* Cirrhosis, chronic active liver disease.
* History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease).
* Any Active systemic infection or history of serious infection within one month.
* Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure , chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases).
* Active tuberculosis
* Malignant hypertension that is difficult to be controlled by oral drugs.
* Known allergy, contraindication or intolerance to the steroids.
* Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception.
* Malignant tumors
* Excessive drinking or drug abuse
* Mental aberrations
* Current or recent (within 30 days) exposure to any other investigational drugs.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Remission of proteinuria (complete or partial) | up to 6 months

SECONDARY OUTCOMES:
Deterioration of renal function (evidenced by a 50% rise from baseline serum creatinine (SCr) levels, or a 25% decline from baseline eGFR levels, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation). | up to 6 months
The longitudinal decline of kidney function(eGFR) | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zongpei Jiang, M.D. & Ph.D., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (6):
- China (6):
  - Department of Nephrology,Dongguan People's Hospital, Dongguan, Guangdong
  - Department of Nephrology, 2nd Affiliated Hospital,Guangzhou Medical University, Guangzhou, Guangdong
  - Department of Nephrology, 6th Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Nephrology,Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Department of Nephrology,1st Affiliated Hospital,Shenzhen University, Shenzhen, Guangdong
  - Department of Nephrology,1st People's Hospital of Zhaoqing, Zhaoqing, Guangdong

REFERENCES:
- [Derived] Liang M, Xiong L, Li A, Zhou J, Huang Y, Huang M, Zhang X, Shi H, Su N, Wei Y, Jiang Z. The effectiveness and safety of corticosteroid therapy for IgA nephropathy with crescents: a prospective, randomized, controlled study. BMC Nephrol. 2022 Jan 21;23(1):40. doi: 10.1186/s12882-022-02661-6. PMID 35062886